CLINICAL TRIAL: NCT04281264
Title: Strength Training in Hypoxia to Improve Bone and Cardiovascular Health of Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Rafael Timón, PhD, Head of research group GAEDAF, University of Extremadura
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: IB18010
Record Dates: First submitted 2020-02-14; First posted 2020-02-24 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Aging Well
Keywords: bone mineral density; healthy aging; resistance training; normobaric hypoxia; cardiovascular health

STUDY DESIGN:
Intervention Model Description: Randomized control trial, in which the experimental sample will be divided into 6 groups where different intervention programs will be performed
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- NorCON (No Intervention): Normoxia Control Group
- HypCON (Active Comparator): Hypoxia Control Group
  Interventions: Behavioral: Passive Hypoxia
- NorCIR (Placebo Comparator): Normoxia Circuit Training with Elastic Bands Group
  Interventions: Behavioral: Normoxia Circuit Training with Elastic Bands
- HypCIR (Experimental): Hypoxia Circuit Training with Elastic Bands Group
  Interventions: Behavioral: Hypoxia Circuit Training with Elastic Bands
- NorVIB (Placebo Comparator): Normoxia Whole-body Vibration Training Group
  Interventions: Behavioral: Normoxia Vibration
- HypVIB (Experimental): Hypoxia Whole-body Vibration Training Group
  Interventions: Behavioral: Hypoxia Vibration

INTERVENTIONS:
Behavioral: Passive Hypoxia — During 30 minutes of session, the participants will perform an intellectual activity while they will be exposed to normobaric hypoxic conditions in a hypoxic chamber (CAT 310, Lousiville, Colorado). They will inspire oxygen fraction (FiO2) set to 16.1% (0.16)
  Arms: HypCON
Behavioral: Normoxia Circuit Training with Elastic Bands — Each training sessions will consist of a circuit training with elastic bands, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit that will be composed by 3 sets of 12-15 repetitions of nine different exercises.
  Subjects will inspire FiO2 of 21.0% (0.21)
  Arms: NorCIR
Behavioral: Hypoxia Circuit Training with Elastic Bands — Each training sessions will consist of a circuit training with elastic bands, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit that will be composed by 3 sets of 12-15 repetitions of nine different exercises.
  Subjects will inspire FiO2 of 21.0% (0.21)
  Arms: HypCIR
Behavioral: Normoxia Vibration — The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles.
  Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1-12 and 45 seconds between 5 repetitions during weeks 12-24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performed on platform.
  Subjects will inspire FiO2 of 21.0% (0.21)
  Arms: NorVIB
Behavioral: Hypoxia Vibration — The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles.
  Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1-12 and 45 seconds between 5 repetitions during weeks 12-24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performance on the platform.
  Participants will inspire a fraction of inspired oxygen (FiO2) of 16.1% (0.16)
  Arms: HypVIB

SUMMARY:
Due to age-related effects, the bone and cardiovascular health are damaged. Physical exercise and in particular the strength training has been proposed as a fundamental tool to these pathologies, especially in the elderly. On the other hand, the use of normobaric hypoxia combined with exercise could have a beneficial synergistic effect on disease prevention and the quality of life of the elderly.

Therefore, the general objective of this project is to analyze the effects of different methods of strength training combined with conditions of normobaric hypoxia on the bone and cardiovascular health of the elderly. This general objective is specified in the following specific objectives:

* To analyze the effects of circuit training with elastic bands on bone mineral density and bone remodelling markers of elderly, under normoxic and normobaric hypoxic conditions.
* To analyze the effects of circuit training with elastic bands on biochemical parameters, inflammatory, endothelial and clinical markers just like cardiovascular risk level of elderly, under normoxic and normobaric hypoxic conditions.
* To analyze the effects of circuit training with elastic bands on body composition and functional capacity of elderly, under normoxic and normobaric hypoxic conditions.
* To analyze the effects of whole-body vibration training on bone mineral density and bone remodelling markers of elderly, under normoxic and normobaric hypoxic conditions.
* To analyze the effects of whole-body vibration training on biochemical parameters, inflammatory, endothelial and clinical markers just like cardiovascular risk level of elderly, under normoxic and normobaric hypoxic conditions.
* To analyze the effects of whole-body vibration training on body composition and functional capacity of elderly, under normoxic and normobaric hypoxic conditions.
* To compare the effects of circuit training with elastic bands versus whole-body vibration training on bone and cardiovascular health of elderly, under normoxic and normobaric hypoxic conditions.
* To value the normobaric hypoxic environment efficacy on bone and cardiovascular health of elderly subjected to circuit training with elastic bands and whole-body vibration training.

We hypothesize that bone and cardiovascular health will improve in the participants subjected to both resistance training, but greater improved may be found when these protocol are combined with normobaric hypoxia.

DETAILED DESCRIPTION:
Participants:

Various associations of pensioners will be contacted as well as the university of seniors of the University of Extremadura to recruit volunteer participants. Total sample size will be 120 people, being this calculated to obtaining a statistical power of 90%, calculated with a margin of error of 5% and a mean difference of 10% in the study variables Design All interventions will be performed during 24 weeks, with a frequency training of 3 days per weeks; sessions will be scheduled with at least one day of rest in between for optimal recovery. All patients were assessed at two time points: at baseline before intervention (Pre) and reassessed 7 days after the last session (Post). Participants will be instructed to continue with their normal daily activities, diet and caloric and calcium intake for the entire duration of the study.

Interventions:

During several times of the session in each intervention, oxygen saturation (SpO2) will be controlled using a finger pulse-oximeter (Konica Minolta, Japan) and heart rate (HR) using a heart rate monitor (Polar team 2, Polar, Finland) to know the physiological challenge posed on the participants during the exposure.

PASSIVE HYPOXIA:

During 30 minutes of session, the participants will be performed an intellectual activity while they will be exposed to normobaric hypoxic conditions in a hypoxic chamber (CAT 310, Lousiville, Colorado). They will inspire oxygen fraction (FiO2) set to 16.1% (0.16) in order to simulate an altitude of 2500m above sea level.

NORMOXIA CIRCUIT TRAINING WITH ELASTIC BANDS Each training sessions will consist of a circuit training, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit that will be composed by 3 sets of 12-15 repetitions of nine different exercises. Six exercises will be performed using elastic resistance bands (ERS; TheraBand®): chest press, row, glute kickbacks, front and side raises, standing bíceps curls and triceps kickbacks. To provide resistance with ERB, elastic bands with resistance ranging from light to very heavy loading (colors: yellow-gold) were used. ERBs were 2 meters, but the actual length used (grip on ERBs and distance to anchor point) was fine tuned for each subject in each exercise to find the correct resistance. When necessary to increase loading, two or more bands were combined. Bands were prestretched and never elongated more than 300% of resting length, as recommended by the manufacturer. Two additional exercise will be developed with kettlebell (KB): squat with 6 kg or increase loading until 10 kg; and hip trust, increase loading with support of a foot alone or with additional loading (KB of 5 or 10 kg). Finally, the subjects will keep a plank position during 15-20 seconds.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. In order to blind subjects to altitude, the system will be run with normoxic airflow into the chamber (up to 1000 l/min) and will produce the same audible noise as in the hypoxic condition. Subjects will inspire FiO2 of 21.0% (0.21) to simulate an altitude of 459 m above sea level. Furthermore, all systems will be covered with fabric to prevent participants from visually identifying the normoxic or hypoxic conditions. FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).

HYPOXIA CIRCUIT TRAINING WITH ELASTIC BANDS Each training sessions will consist of a circuit training, where different muscle groups will be involved (pectoral, shoulders, back, arms, thighs, legs and abdominals). Duration of the session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the sessions. Main section of the sessions will be a circuit, that will be composed by 3 sets of 12-15 repetitions of nine different exercises. Six exercises will be performed using elastic resistance bands (ERS; TheraBand®): chest press, row, glute kickbacks, front and side raises, standing bíceps curls and triceps kickbacks. To provide resistance with ERB, elastic bands with resistance ranging from light to very heavy loading (colors: yellow-gold) were used. ERBs were 2 meters, but the actual length used (grip on ERBs and distance to anchor point) was fine tuned for each subject in each exercise to find the correct resistance. When necessary to increase loading, two or more bands were combined. Bands were prestretched and never elongated more than 300% of resting length, as recommended by the manufacturer. Two additional exercise will be developed with kettlebell (KB): squat with 6 kg or increase loading until 10 kg; and hip trust, increase loading with support of a foot alone or with additional loading (KB of 5 or 10 kg). Finally, the subjects will keep a plank position during 15-20 seconds Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. Participants will inspire a fraction of inspired oxygen (FiO2) of 16.1% (0.16) to simulate an altitude of 2500 m above sea level; FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).

NORMOXIA WHOLE-BODY VIBRATION The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the session.

Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1-12 and 45 seconds between 5 repetitions during weeks 12-24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performance, with the soles of both feet remained in contact with the platform:

1. Stand with feet side-by-side on the board, which produced lateral oscillations of the whole body. During the vibration training sessions, the subjects will be barefoot to eliminate any damping of the vibration caused by footwear. The angle of flexion of the knees during the vibration exercise will be set at 60°.
2. Begin with the feet placed perpendicular to the midline axis of the platform, with a foot positioned slightly ahead of the other foot. Lift the toes of the one foot and the heel of the other foot 4 mm above the surface of the platform. Bend the knees and maintain a 45°knee angle. Keep the back and head straight. Alternate legs.
3. Front foot 4 mm above the surface of the platform and back foot on ground, front knee angle 90°. Alternate legs
4. Lay down on the ground, with the knees bent and feet flat on the platform. Keep the arms at your side with your palms down. Lift the hips off the ground until the knees, hips and shoulders form a straight line. Hold your bridged position.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. In order to blind subjects to altitude, the system will be run with normoxic airflow into the chamber (up to 1000 l/min) and will produce the same audible noise as in the hypoxic condition. Subjects will inspire FiO2 of 21.0% (0.21) to simulate an altitude of 459 m above sea level. Furthermore, all systems will be covered with fabric to prevent participants from visually identifying the normoxic or hypoxic conditions. FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).

HYPOXIA WHOLE-BODY VIBRATION The subjects will perform dynamic and static vibration exercise provide by a commercially available device (Galileo 2000, Novotec GmbH, Pforzheim, Alemania). The duration of the WBV session will be about 30 minutes, which will include 10 minutes warm-up consisting of slight movements, and 5 minutes of static stretching for the muscles at the end of the session.

Repetitions of 30 seconds with a frequency of 18.5 Hz will be performed. The rest interval will be 60 seconds between 4 repetitions during weeks 1-12 and 45 seconds between 5 repetitions during weeks 12-24. The vertical amplitude of WBV was set at 2.5 mm. Four stance will be performance, with the soles of both feet remained in contact with the platform:

1. Stand with feet side-by-side on the board, which produced lateral oscillations of the whole body. During the vibration training sessions, the subjects will be barefoot to eliminate any damping of the vibration caused by footwear. The angle of flexion of the knees during the vibration exercise will be set at 60°.
2. Begin with the feet placed perpendicular to the midline axis of the platform, with a foot positioned slightly ahead of the other foot. Lift the toes of the one-foot and the heel of the other foot 4 mm above the surface of the platform. Bend the knees and maintain a 45°knee angle. Keep the back and head straight. Alternate legs.
3. Front foot 4 mm above the surface of the platform and back foot on ground, front knee angle 90°. Alternate legs
4. Lay down on the ground, with the knees bent and feet flat on the platform. Keep the arms at your side with your palms down. Lift the hips off the ground until the knees, hips and shoulders form a straight line. Hold your bridged position.

Training will take place in a hypoxia chamber (CAT 310, Lousiville, Colorado, United States) will place in the laboratory. Participants will inspire a fraction of inspired oxygen (FiO2) of 16.1% (0.16) to simulate an altitude of 2500 m above sea level; FiO2 will be controlled regularly with an electronic device (HANDIC,Maxtec, Salt Lake City, Utah, United States).

Statistical Analysis Statistical analyses will be performed using the statistical analysis package SPSS v.20 (IBM, New York, United States). Data will be expressed as median and standard deviation. Kolmogorov-Smirnov tests will be conducted to show the distribution of the studied variables and Levene's test for homogeneity of variance. Repeated measure ANOVA will be used to compare the response of each variable, considering the sex and age as covariate. The p < 0.05 criterion was used for establishing statistical significance. Effect size (Cohen, 1992) will be also calculated for all variables, considering the magnitude of change as small (0.2), moderate (0.5) or large (0.8).

ELIGIBILITY:
Inclusion Criteria:

1. women and men aged 65 years or older
2. no current medical condition not compatible with planned exercise
3. free of illness or medication potentially affecting the bone and cardiovascular system
4. estimated daily calcium intake of 1200-2000 mg/day
5. consumption of no more than two alcoholic beverages per day.

Exclusion Criteria:

1. participation in any other type of intervention based on physical exercise in the last 6 months in order to avoid interactions with the previous practice
2. subjects have been above 1500 m during the last 3 months
3. contra indications for whole-body vibration training: severe cardiovascular diseases, ocular diseases that affect the retina, neuromuscular and heart diseases, stroke, implant, bypass, stent, arthritis and other joint disease or epilepsy

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Life Quality at 24 weeks | Through study completion, an average of 24 weeks
  SF-36 questionnaire will be used to know the life quality
Change from Baseline Risk of Fall at 24 weeks | Through study completion, an average of 24 weeks
  Risk of fall will be evaluated through Fall Efficacy Scale-International (FES-I)
Change from Baseline Blood Pressure at 24 weeks | Through study completion, an average of 24 weeks
  Blood pressure (mmHg) will be measured with sphygmomanometer
Change from Baseline Cardiovascular Evaluation at 24 weeks | Through study completion, an average of 24 weeks
  Arm-ankle index and pulse wave velocity will be measured using ultrasound Doppler technique
Change from Baseline Cardiovascular Risk at 24 weeks | Through study completion, an average of 24 weeks
  Based on the following factors: age, sex, smoking, total cholesterol, HDL cholesterol, systolic blood pressure and diabetes, cardiovascular risk will be determined. This method was already described in the FRESCO study
Change from Baseline Weight at 24 weeks | Through study completion, an average of 24 weeks
  Weight (kilograms) will measure following standard procedures
Change from Baseline Height at 24 weeks | Through study completion, an average of 24 weeks
  Height (meters) will measure following standard procedures
Change from Baseline Body Mass Index at 24 weeks | Through study completion, an average of 24 weeks
  Weight and Height will be combined to report body mass index (BMI) in kg/m^2
Change from Baseline Waist-Hip Ratio at 24 weeks | Through study completion, an average of 24 weeks
  Waist and hip diameter (centimeters) will be combined to report Waist-Hip Ratio
Change from Baseline Body Composition at 24 weeks | Through study completion, an average of 24 weeks
  Body composition variables such as percentage fat and lean fat mass (percentage) will be obtain using dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States).
Change from Baseline Bone Mineral Density at 24 weeks | Through study completion, an average of 24 weeks
  Bone mineral density (g/cm-2) of whole body and proximal femur region will be calculated from obtained data of dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States)
Change from Baseline Osteoporosis/Osteopenia Prevalence at 24 weeks | Through study completion, an average of 24 weeks
  T-score of whole body and proximal femur region will be calculated from obtained data of dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States)
Change from Baseline Bone Mineral Content at 24 weeks | Through study completion, an average of 24 weeks
  Bone mineral content (g) of whole body and proximal femur region will be calculated from obtained data of dual-energy X-ray absorptiometry (DXA,Norland Excell Plus; Norland Inc., Fort Atkinson, United States)
Change from Baseline Biochemical Parameters at 24 weeks | Through study completion, an average of 24 weeks
  Standard biochemical analysis (HDL, LDL and Total Cholesterol, Triglycerides and Glucose in mg/dL) will be obtained of blood samples, through a clinical chemistry analyzer (Spotchem, Arkray Factory, Germany)
Change from Baseline Bone Remodelling Markers at 24 weeks | Through study completion, an average of 24 weeks
  Bone remodelling (VEGF and SDF-1 in mg/dL) markers will be analyzed by ELISA technique.
Change from Baseline Inflammatory Markers at 24 weeks | Through study completion, an average of 24 weeks
  Inflammatory (C-reactive protein, IL-2, IL-4, IL-6 and TNFa in mg/dL) markers will be analyzed by ELISA technique.
Change from Baseline Endothelial Markers at 24 weeks | Through study completion, an average of 24 weeks
  Endothelial (ICAM-1 and VCAM-1 in mg/dL) markers will be analyzed by ELISA technique.
Change from Baseline Lower Limb Strength at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Lower limb strength will be tested by Chair stand Test (repetitions)
Change from Baseline Upper Limb Strength at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Upper limb strength will be tested by Arm curl Test (repetitions)
Change from Baseline Lower Limb Flexibility at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Lower limb flexibility will be tested by Chair sit and reach Test (centimeters)
Change from Baseline Upper Limb Flexibility at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Upper limb flexibility will be tested by Back scratch Test (centimeters)
Change from Baseline Endurance at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Endurance will be tested by 6 min. walk Test (meters)
Change from Baseline Agility at 24 weeks | Through study completion, an average of 24 weeks
  Senior Fitness Test battery will be used to know of physical condition of elderly. Agility will be tested by 8ft Up and Go Test (seconds).
Change from Baseline Core muscle strength at 24 weeks | Through study completion, an average of 24 weeks
  Core muscle strength will be tested by plank test (seconds)
Change from Baseline Grip strength at 24 weeks | Through study completion, an average of 24 weeks
  Grip strength will be tested using an Handgrip (kilograms)
Change from Baseline Balance at 24 weeks | Through study completion, an average of 24 weeks
  Balance will be tested by single leg stance test (seconds)

SECONDARY OUTCOMES:
Socio-Demographic Data | Baseline
  A general questionnaire was administered to collect medical and demographic data to check the inclusion/exclusion criteria.
Change from Baseline Calcium Intake at 24 weeks | Through study completion, an average of 24 weeks
  Calcium intake (mg/day) will be estimated using a food frequency questionnaire
Change from Baseline Physical Activity Level at 24 weeks | Through study completion, an average of 24 weeks
  The bone-specific physical activity questionnaire (B-PAQ; score) will be used to assess the physical activity level of the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Sport Science Faculty. University of Extremadura, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhella PS, Hastings JL, Fujimoto N, Shibata S, Carrick-Ranson G, Palmer MD, Boyd KN, Adams-Huet B, Levine BD. Impact of lifelong exercise "dose" on left ventricular compliance and distensibility. J Am Coll Cardiol. 2014 Sep 23;64(12):1257-66. doi: 10.1016/j.jacc.2014.03.062. PMID 25236519
- [Background] Bliuc D, Nguyen ND, Milch VE, Nguyen TV, Eisman JA, Center JR. Mortality risk associated with low-trauma osteoporotic fracture and subsequent fracture in men and women. JAMA. 2009 Feb 4;301(5):513-21. doi: 10.1001/jama.2009.50. PMID 19190316
- [Background] Bogaerts A, Delecluse C, Boonen S, Claessens AL, Milisen K, Verschueren SM. Changes in balance, functional performance and fall risk following whole body vibration training and vitamin D supplementation in institutionalized elderly women. A 6 month randomized controlled trial. Gait Posture. 2011 Mar;33(3):466-72. doi: 10.1016/j.gaitpost.2010.12.027. Epub 2011 Jan 20. PMID 21256028
- [Background] Buckinx F, Beaudart C, Maquet D, Demonceau M, Crielaard JM, Reginster JY, Bruyere O. Evaluation of the impact of 6-month training by whole body vibration on the risk of falls among nursing home residents, observed over a 12-month period: a single blind, randomized controlled trial. Aging Clin Exp Res. 2014 Aug;26(4):369-76. doi: 10.1007/s40520-014-0197-z. Epub 2014 Jan 28. PMID 24469903
- [Background] Burghardt AJ, Buie HR, Laib A, Majumdar S, Boyd SK. Reproducibility of direct quantitative measures of cortical bone microarchitecture of the distal radius and tibia by HR-pQCT. Bone. 2010 Sep;47(3):519-28. doi: 10.1016/j.bone.2010.05.034. Epub 2010 May 31. PMID 20561906
- [Background] Celis-Morales CA, Welsh P, Lyall DM, Steell L, Petermann F, Anderson J, Iliodromiti S, Sillars A, Graham N, Mackay DF, Pell JP, Gill JMR, Sattar N, Gray SR. Associations of grip strength with cardiovascular, respiratory, and cancer outcomes and all cause mortality: prospective cohort study of half a million UK Biobank participants. BMJ. 2018 May 8;361:k1651. doi: 10.1136/bmj.k1651. PMID 29739772
- [Background] Cenzer IS, Tang V, Boscardin WJ, Smith AK, Ritchie C, Wallhagen MI, Espaldon R, Covinsky KE. One-Year Mortality After Hip Fracture: Development and Validation of a Prognostic Index. J Am Geriatr Soc. 2016 Sep;64(9):1863-8. doi: 10.1111/jgs.14237. Epub 2016 Jun 13. PMID 27295578
- [Background] Chan DA, Sutphin PD, Denko NC, Giaccia AJ. Role of prolyl hydroxylation in oncogenically stabilized hypoxia-inducible factor-1alpha. J Biol Chem. 2002 Oct 18;277(42):40112-7. doi: 10.1074/jbc.M206922200. Epub 2002 Aug 16. PMID 12186875
- [Background] Cummings SR, Melton LJ. Epidemiology and outcomes of osteoporotic fractures. Lancet. 2002 May 18;359(9319):1761-7. doi: 10.1016/S0140-6736(02)08657-9. PMID 12049882
- [Background] Delecluse C, Roelants M, Verschueren S. Strength increase after whole-body vibration compared with resistance training. Med Sci Sports Exerc. 2003 Jun;35(6):1033-41. doi: 10.1249/01.MSS.0000069752.96438.B0. PMID 12783053
- [Background] Dreimuller N, Schlicht KF, Wagner S, Peetz D, Borysenko L, Hiemke C, Lieb K, Tadic A. Early reactions of brain-derived neurotrophic factor in plasma (pBDNF) and outcome to acute antidepressant treatment in patients with Major Depression. Neuropharmacology. 2012 Jan;62(1):264-9. doi: 10.1016/j.neuropharm.2011.07.017. Epub 2011 Jul 22. PMID 21803060
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Fratini A, Bonci T, Bull AM. Whole Body Vibration Treatments in Postmenopausal Women Can Improve Bone Mineral Density: Results of a Stimulus Focussed Meta-Analysis. PLoS One. 2016 Dec 1;11(12):e0166774. doi: 10.1371/journal.pone.0166774. eCollection 2016. PMID 27907000
- [Background] Gianoudis J, Bailey CA, Ebeling PR, Nowson CA, Sanders KM, Hill K, Daly RM. Effects of a targeted multimodal exercise program incorporating high-speed power training on falls and fracture risk factors in older adults: a community-based randomized controlled trial. J Bone Miner Res. 2014 Jan;29(1):182-91. doi: 10.1002/jbmr.2014. PMID 23775701
- [Background] Gonzalez-Aguero A, Vicente-Rodriguez G, Gomez-Cabello A, Casajus JA. Cortical and trabecular bone at the radius and tibia in male and female adolescents with Down syndrome: a peripheral quantitative computed tomography (pQCT) study. Osteoporos Int. 2013 Mar;24(3):1035-44. doi: 10.1007/s00198-012-2041-7. Epub 2012 Jun 9. PMID 22684498
- [Background] Goudarzian M, Ghavi S, Shariat A, Shirvani H, Rahimi M. Effects of whole body vibration training and mental training on mobility, neuromuscular performance, and muscle strength in older men. J Exerc Rehabil. 2017 Oct 30;13(5):573-580. doi: 10.12965/jer.1735024.512. eCollection 2017 Oct. PMID 29114533
- [Background] Graham I, Atar D, Borch-Johnsen K, Boysen G, Burell G, Cifkova R, Dallongeville J, De Backer G, Ebrahim S, Gjelsvik B, Herrmann-Lingen C, Hoes A, Humphries S, Knapton M, Perk J, Priori SG, Pyorala K, Reiner Z, Ruilope L, Sans-Menendez S, Op Reimer WS, Weissberg P, Wood D, Yarnell J, Zamorano JL, Walma E, Fitzgerald T, Cooney MT, Dudina A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Funck-Brentano C, Filippatos G, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Altiner A, Bonora E, Durrington PN, Fagard R, Giampaoli S, Hemingway H, Hakansson J, Kjeldsen SE, Larsen mL, Mancia G, Manolis AJ, Orth-Gomer K, Pedersen T, Rayner M, Ryden L, Sammut M, Schneiderman N, Stalenhoef AF, Tokgozoglu L, Wiklund O, Zampelas A; European Society of Cardiology (ESC); European Association for Cardiovascular Prevention and Rehabilitation (EACPR); Council on Cardiovascular Nursing; European Association for Study of Diabetes (EASD); International Diabetes Federation Europe (IDF-Europe); European Stroke Initiative (EUSI); Society of Behavioural Medicine (ISBM); European Society of Hypertension (ESH); WONCA Europe (European Society of General Practice/Family Medicine); European Heart Network (EHN); European Atherosclerosis Society (EAS). European guidelines on cardiovascular disease prevention in clinical practice: full text. Fourth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts). Eur J Cardiovasc Prev Rehabil. 2007 Sep;14 Suppl 2:S1-113. doi: 10.1097/01.hjr.0000277983.23934.c9. No abstract available. PMID 17726407
- [Background] Guner I, Uzun DD, Yaman MO, Genc H, Gelisgen R, Korkmaz GG, Hallac M, Yelmen N, Sahin G, Karter Y, Simsek G. The effect of chronic long-term intermittent hypobaric hypoxia on bone mineral density in rats: role of nitric oxide. Biol Trace Elem Res. 2013 Aug;154(2):262-7. doi: 10.1007/s12011-013-9722-8. Epub 2013 Jun 16. PMID 23771686
- [Background] Hinton PS, Nigh P, Thyfault J. Effectiveness of resistance training or jumping-exercise to increase bone mineral density in men with low bone mass: A 12-month randomized, clinical trial. Bone. 2015 Oct;79:203-12. doi: 10.1016/j.bone.2015.06.008. Epub 2015 Jun 16. PMID 26092649
- [Background] Inness MW, Billaut F, Walker EJ, Petersen AC, Sweeting AJ, Aughey RJ. Heavy Resistance Training in Hypoxia Enhances 1RM Squat Performance. Front Physiol. 2016 Nov 3;7:502. doi: 10.3389/fphys.2016.00502. eCollection 2016. PMID 27857693
- [Background] Johnell O, Kanis J. Epidemiology of osteoporotic fractures. Osteoporos Int. 2005 Mar;16 Suppl 2:S3-7. doi: 10.1007/s00198-004-1702-6. Epub 2004 Sep 8. PMID 15365697
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- [Background] Kawanabe K, Kawashima A, Sashimoto I, Takeda T, Sato Y, Iwamoto J. Effect of whole-body vibration exercise and muscle strengthening, balance, and walking exercises on walking ability in the elderly. Keio J Med. 2007 Mar;56(1):28-33. doi: 10.2302/kjm.56.28. PMID 17392595
- [Background] Kon M, Ohiwa N, Honda A, Matsubayashi T, Ikeda T, Akimoto T, Suzuki Y, Hirano Y, Russell AP. Effects of systemic hypoxia on human muscular adaptations to resistance exercise training. Physiol Rep. 2014 Jun 6;2(6):e12033. doi: 10.14814/phy2.12033. Print 2014 Jun 1. PMID 24907297
- [Background] Kraemer WJ, Ratamess NA, French DN. Resistance training for health and performance. Curr Sports Med Rep. 2002 Jun;1(3):165-71. doi: 10.1249/00149619-200206000-00007. PMID 12831709
- [Background] McMillan LB, Zengin A, Ebeling PR, Scott D. Prescribing Physical Activity for the Prevention and Treatment of Osteoporosis in Older Adults. Healthcare (Basel). 2017 Nov 6;5(4):85. doi: 10.3390/healthcare5040085. PMID 29113119
- [Background] Mikhael M, Orr R, Amsen F, Greene D, Singh MA. Effect of standing posture during whole body vibration training on muscle morphology and function in older adults: a randomised controlled trial. BMC Geriatr. 2010 Oct 15;10:74. doi: 10.1186/1471-2318-10-74. PMID 20946685
- [Background] Navarrete-Opazo A, Mitchell GS. Therapeutic potential of intermittent hypoxia: a matter of dose. Am J Physiol Regul Integr Comp Physiol. 2014 Nov 15;307(10):R1181-97. doi: 10.1152/ajpregu.00208.2014. Epub 2014 Sep 17. PMID 25231353
- [Background] Niino N, Tsuzuku S, Ando F, Shimokata H. Frequencies and circumstances of falls in the National Institute for Longevity Sciences, Longitudinal Study of Aging (NILS-LSA). J Epidemiol. 2000 Apr;10(1 Suppl):S90-4. doi: 10.2188/jea.10.1sup_90. PMID 10835834
- [Background] Papa EV, Foreman KB, Dibble LE. Effects of age and acute muscle fatigue on reactive postural control in healthy adults. Clin Biomech (Bristol). 2015 Dec;30(10):1108-13. doi: 10.1016/j.clinbiomech.2015.08.017. Epub 2015 Sep 2. PMID 26351001
- [Background] Papa EV, Garg H, Dibble LE. Acute effects of muscle fatigue on anticipatory and reactive postural control in older individuals: a systematic review of the evidence. J Geriatr Phys Ther. 2015 Jan-Mar;38(1):40-8. doi: 10.1519/JPT.0000000000000026. PMID 24978932
- [Background] Rubin C, Recker R, Cullen D, Ryaby J, McCabe J, McLeod K. Prevention of postmenopausal bone loss by a low-magnitude, high-frequency mechanical stimuli: a clinical trial assessing compliance, efficacy, and safety. J Bone Miner Res. 2004 Mar;19(3):343-51. doi: 10.1359/JBMR.0301251. Epub 2003 Dec 22. PMID 15040821
- [Background] Pouyssegur J, Dayan F, Mazure NM. Hypoxia signalling in cancer and approaches to enforce tumour regression. Nature. 2006 May 25;441(7092):437-43. doi: 10.1038/nature04871. PMID 16724055
- [Background] Sallis R. Exercise is medicine: a call to action for physicians to assess and prescribe exercise. Phys Sportsmed. 2015 Feb;43(1):22-6. doi: 10.1080/00913847.2015.1001938. PMID 25684558
- [Background] Schega L, Peter B, Torpel A, Mutschler H, Isermann B, Hamacher D. Effects of intermittent hypoxia on cognitive performance and quality of life in elderly adults: a pilot study. Gerontology. 2013;59(4):316-23. doi: 10.1159/000350927. Epub 2013 May 3. PMID 23652274
- [Background] Scott BR, Slattery KM, Sculley DV, Dascombe BJ. Hypoxia and resistance exercise: a comparison of localized and systemic methods. Sports Med. 2014 Aug;44(8):1037-54. doi: 10.1007/s40279-014-0177-7. PMID 24715613
- [Background] Shaw BS, Shaw I, Mamen A. Contrasting effects in anthropometric measures of total fatness and abdominal fat mass following endurance and concurrent endurance and resistance training. J Sports Med Phys Fitness. 2010 Jun;50(2):207-13. PMID 20585300
- [Background] Shaw I, Shaw BS, Brown GA, Cilliers JF. Concurrent resistance and aerobic training as protection against heart disease. Cardiovasc J Afr. 2010 Jul-Aug;21(4):196-9. PMID 20838717
- [Background] Sipila S, Elorinne M, Alen M, Suominen H, Kovanen V. Effects of strength and endurance training on muscle fibre characteristics in elderly women. Clin Physiol. 1997 Sep;17(5):459-74. doi: 10.1046/j.1365-2281.1997.05050.x. PMID 9347195
- [Background] Swanson CM, Shea SA, Stone KL, Cauley JA, Rosen CJ, Redline S, Karsenty G, Orwoll ES. Obstructive sleep apnea and metabolic bone disease: insights into the relationship between bone and sleep. J Bone Miner Res. 2015 Feb;30(2):199-211. doi: 10.1002/jbmr.2446. PMID 25639209
- [Background] Tosteson AN, Gottlieb DJ, Radley DC, Fisher ES, Melton LJ 3rd. Excess mortality following hip fracture: the role of underlying health status. Osteoporos Int. 2007 Nov;18(11):1463-72. doi: 10.1007/s00198-007-0429-6. Epub 2007 Aug 29. PMID 17726622
- [Background] von Friesendorff M, McGuigan FE, Wizert A, Rogmark C, Holmberg AH, Woolf AD, Akesson K. Hip fracture, mortality risk, and cause of death over two decades. Osteoporos Int. 2016 Oct;27(10):2945-53. doi: 10.1007/s00198-016-3616-5. Epub 2016 May 12. PMID 27172936
- [Background] Watson SL, Weeks BK, Weis LJ, Horan SA, Beck BR. Heavy resistance training is safe and improves bone, function, and stature in postmenopausal women with low to very low bone mass: novel early findings from the LIFTMOR trial. Osteoporos Int. 2015 Dec;26(12):2889-94. doi: 10.1007/s00198-015-3263-2. Epub 2015 Aug 5. PMID 26243363
- [Background] Westcott WL. Resistance training is medicine: effects of strength training on health. Curr Sports Med Rep. 2012 Jul-Aug;11(4):209-16. doi: 10.1249/JSR.0b013e31825dabb8. PMID 22777332
- [Background] Williams AD, Almond J, Ahuja KD, Beard DC, Robertson IK, Ball MJ. Cardiovascular and metabolic effects of community based resistance training in an older population. J Sci Med Sport. 2011 Jul;14(4):331-7. doi: 10.1016/j.jsams.2011.02.011. Epub 2011 Mar 26. PMID 21441068
- [Background] Zaki ME. Effects of whole body vibration and resistance training on bone mineral density and anthropometry in obese postmenopausal women. J Osteoporos. 2014;2014:702589. doi: 10.1155/2014/702589. Epub 2014 Jun 18. PMID 25136473
- [Background] Zhang L, Weng C, Liu M, Wang Q, Liu L, He Y. Effect of whole-body vibration exercise on mobility, balance ability and general health status in frail elderly patients: a pilot randomized controlled trial. Clin Rehabil. 2014 Jan;28(1):59-68. doi: 10.1177/0269215513492162. Epub 2013 Jul 17. PMID 23864514
- [Background] Zhao R, Zhao M, Xu Z. The effects of differing resistance training modes on the preservation of bone mineral density in postmenopausal women: a meta-analysis. Osteoporos Int. 2015 May;26(5):1605-18. doi: 10.1007/s00198-015-3034-0. Epub 2015 Jan 21. PMID 25603795
- [Background] Zuo C, Huang Y, Bajis R, Sahih M, Li YP, Dai K, Zhang X. Osteoblastogenesis regulation signals in bone remodeling. Osteoporos Int. 2012 Jun;23(6):1653-63. doi: 10.1007/s00198-012-1909-x. PMID 22290242
- [Derived] Timon R, Gonzalez-Custodio A, Gusi N, Olcina G. Effects of intermittent hypoxia and whole-body vibration training on health-related outcomes in older adults. Aging Clin Exp Res. 2024 Jan 27;36(1):6. doi: 10.1007/s40520-023-02655-w. PMID 38280022
- [Derived] Camacho-Cardenosa A, Camacho-Cardenosa M, Martinez-Guardado I, Leal A, Andrada JMV, Timon R. Resistance circuit training combined with hypoxia stimulates bone system of older adults: A randomized trial. Exp Gerontol. 2022 Nov;169:111983. doi: 10.1016/j.exger.2022.111983. Epub 2022 Oct 13. PMID 36243220
- [Derived] Timon R, Camacho-Cardenosa M, Gonzalez-Custodio A, Olcina G, Gusi N, Camacho-Cardenosa A. Effect of hypoxic conditioning on functional fitness, balance and fear of falling in healthy older adults: a randomized controlled trial. Eur Rev Aging Phys Act. 2021 Dec 1;18(1):25. doi: 10.1186/s11556-021-00279-5. PMID 34852758
- [Derived] Timon R, Martinez-Guardado I, Camacho-Cardenosa A, Villa-Andrada JM, Olcina G, Camacho-Cardenosa M. Effect of intermittent hypoxic conditioning on inflammatory biomarkers in older adults. Exp Gerontol. 2021 Sep;152:111478. doi: 10.1016/j.exger.2021.111478. Epub 2021 Jul 10. PMID 34256114

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04281264/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT04281264/ICF_001.pdf